CLINICAL TRIAL: NCT02481154
Title: A Phase 1, Multicenter, Open-Label, Dose-Escalation and Expansion, Safety, Pharmacokinetic, Pharmacodynamic, and Clinical Activity Study of Orally Administered AG-881 in Patients With Advanced Solid Tumors, Including Gliomas, With an IDH1 and/or IDH2 Mutation
Brief Title: Study of Orally Administered AG-881 in Patients With Advanced Solid Tumors, Including Gliomas, With an IDH1 and/or IDH2 Mutation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG881-C-002
Record Dates: First submitted 2015-06-16; First posted 2015-06-25 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Glioma
Keywords: Glioma; IDH1; IDH2; Dual Mutation; AG-881
MeSH Terms: conditions — Glioma

ARMS (1):
- AG881 (Experimental): AG-881 administered continuously as a single agent dosed orally on Days 1 to 28 of a 28-day cycle. Patients may continue treatment with AG-881 until disease progression, development of other unacceptable toxicity or Investigator discretion
  Interventions: Drug: AG881

INTERVENTIONS:
Drug: AG881 — AG-881 administered continuously as a single agent dosed orally on Days 1 to 28 of a 28-day cycle. Patients may continue treatment with AG-881 until disease progression or development of other unacceptable toxicity

SUMMARY:
This study evaluates the safety, pharmacokinetics, pharmacodynamics and clinical activity of AG-881 in Gliomas, that harbor an IDH1 and/or IDH2 mutation.

DETAILED DESCRIPTION:
The purpose of this Phase I, multicenter study is to evaluate the safety, pharmacokinetics, pharmacodynamics and clinical activity of AG-881 in gliomas, that harbor an IDH1and/or IDH2 mutation. The first portion of the study is a dose escalation phase where cohorts of patients will receive ascending oral doses of AG-881 to determine the maximum tolerated dose (MTD) and/or the recommended Phase II dose. The second portion of the study is a dose expansion phase where patients will receive AG-881 to further evaluate the safety, tolerability, and clinical activity of the recommended Phase II dose. The anticipated time on study treatment is until disease progression, unacceptable toxicity occurs or the patient is removed at the discretion of the investigator

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥18 years of age
* Patient must have histologically or cytologically confirmed solid tumor, including glioma, with documented IDH1 and/or IDH2 gene-mutation. Patients in the dose escalation phase must have disease that has recurred or progressed following standard therapy and/or therapy with an inhibitor of mutant IDH1 and/or IDH2, or that has not responded to this therapy. Patients in the expansion phase may have previously untreated disease
* Patient must have evaluable disease by RECIST v1.1 for patients without glioma or by RANO or RANO LGG criteria for patients with glioma
* Patients with glioma must have a baseline brain MRI scan
* Patient must have archived primary tumor biopsies or surgical specimens, or biopsies of recurrent or metastatic samples
* Patient must be amenable to serial peripheral blood sampling, urine sampling, and tumor biopsies during the study
* Patient must be able to understand and willing to sign an informed consent
* Patient must have ECOG PS of 0 to 2
* Patient must have expected survival of ≥3 months
* Patient must have adequate bone marrow function as evidenced by absolute neutrophil count ≥1.5 ×10^9/L; hemoglobin >9 g/dL (Patients are allowed to be transfused to this level); platelets ≥75 × 10^9/L
* Patient must have adequate hepatic function as evidenced by: Serum total bilirubin ≤1.5 × upper limit of normal (ULN), unless considered due to Gilbert's disease or disease involvement; Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤2.5 × ULN. For patients with bone metastases and/or suspected disease-related liver or biliary involvement, AST, ALT and ALP must be ≤5 × ULN
* Patient must have adequate renal function as evidenced by: Serum creatinine ≤2.0 × ULN or Creatinine clearance >40 mL/min based on the Cockroft-Gault glomerular filtration rate (GFR) estimated: (140-Age) x (weight in kg) x (0.85 if female)/72 x serum creatinine
* Patient must be recovered from any clinically relevant toxic effects of any prior surgery, radiotherapy, or other therapy intended for the treatment of cancer
* Female patients with reproductive potential must have a negative serum pregnancy test within 7 days prior to first study drug administration. Patients with reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy or tubal occlusion or who have not experienced natural menopause (i.e., who have not menstruated at all) for at least 24 consecutive months (i.e., have had menses at any time in the preceding 24 consecutive months). Women with reproductive potential as well as fertile men and their partners who are female with reproductive potential must agree to abstain from sexual intercourse or to use two highly effective forms of contraception from the time of giving informed consent, during the study, and for 90 days (females and males) following the last dose of AG 881

Exclusion Criteria:

* Patients who received systemic anticancer therapy or radiotherapy <21 days prior to their first day of study drug administration
* Patients who received an investigational agent (including AG-120 or AG-221) <14 days prior to their first day of study drug administration. In addition, the first dose of AG-881 should not occur before a period ≥5 half-lives of the investigational agent (other than AG-120 or AG-221) has elapsed.
* Patients with gliomas who have had prior treatment with bevacizumab (Avastin) are excluded
* Patients who are pregnant or breast feeding
* Patients with an active severe infection that required anti-infective therapy or with an unexplained fever >38.5°C during screening visits or on their first day of study drug administration (at the discretion of the Investigator, patients with tumor fever may be enrolled)
* Patients with New York Heart Association (NYHA) Class III or IV congestive heart failure or LVEF <40% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan obtained within approximately 28 days of C1D1
* Patients with a history of myocardial infarction within the 6 months prior to screening
* Patients with known unstable or uncontrolled angina pectoris
* Patients with a known history of severe and/or uncontrolled ventricular arrhythmias
* Patients with QTc interval ≥450 msec or with other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome)
* Patients taking medications that are known to prolong the QT interval unless they can be transferred to other medications within ≥5 half-lives prior to dosing, or unless the medications can be properly monitored during the study.
* Patients with known infection with human immunodeficiency virus (HIV) or active hepatitis B or C
* Patients with known dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally
* Patients with brain metastases that are untreated, symptomatic, or require therapy to control symptoms; or any radiation, surgery, or other therapy, including those used to control symptoms, within 1 month of first dose
* Glioma patients with evidence of intracranial or intratumoral hemorrhage either by MRI or CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Safety/Tolerability; incidence of adverse events | Up to 26 weeks, on average
Maximum Tolerated Dose and/or the recommended Phase II dose of AG881 in patients with advance solid tumors, including gliomas | Up to 26 weeks, on average

SECONDARY OUTCOMES:
Pharmacokinetic profiles including max concentration (Cmax), time to maximum concentration (Tmax), AUC, and elimination half-life | Up to 26 weeks, on average
Pharmacodynamic levels of AG-881 | Up to 26 weeks, on average
Pharmacodynamic levels of 2-HG | Up to 26 weeks, on average
Clinical Activity according to RECIST v 1.1 (2009) for patients with solid tumors, by RANO (2010) criteria for patients with glioma | Up to 26 weeks, on average

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - UCLA Oncology Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Derived] Mellinghoff IK, Penas-Prado M, Peters KB, Burris HA 3rd, Maher EA, Janku F, Cote GM, de la Fuente MI, Clarke JL, Ellingson BM, Chun S, Young RJ, Liu H, Choe S, Lu M, Le K, Hassan I, Steelman L, Pandya SS, Cloughesy TF, Wen PY. Vorasidenib, a Dual Inhibitor of Mutant IDH1/2, in Recurrent or Progressive Glioma; Results of a First-in-Human Phase I Trial. Clin Cancer Res. 2021 Aug 15;27(16):4491-4499. doi: 10.1158/1078-0432.CCR-21-0611. Epub 2021 Jun 2. PMID 34078652
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/